CLINICAL TRIAL: NCT04290624
Title: A Randomized, Controlled Clinical Study to Evaluate the Efficacy of a Range of Dental/Denture Products for Improved Oral Health, Compared to Existing Oral Hygiene, in a Population of Partial Denture Wearers With Generalized Mild-moderate Plaque-induced Gingivitis
Brief Title: A Clinical Study to Evaluate the Efficacy of a Range of Dental/Denture Products for Improved Oral Health in Partial Denture Wearers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 212401; 212401 (Other: GlaxoSmithKline)
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-02

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will be instructed to use a dentifrice containing 0.454 percent (%) weight by weight (w/w) Stannous fluoride, COREGA denture foaming cleanser and mouth rinse containing 90 parts per million (ppm) sodium fluoride. Participants will brush with a strip of the dentifrice (full brush head) applied to the full length of the toothbrush head for 2 minutes followed by 2 pumps of denture cleanser foam brushed onto removable partial denture (RPD) for 90 seconds and 10 milliliter (ml) of mouth rinse for swished around the mouth for 1 minute. Participants will apply all these products twice daily (morning and evening) for 12 weeks.
  Interventions: Other: Experimental Dentifrice: Stannous Fluoride; Device: COREGA Denture Foaming Cleanser; Other: Mouth rinse: Sodium Fluoride
- Reference Group (No Intervention): Participants will not be supplied any products and will continue with their existing dental/denture hygiene practices and should not make changes to either their established habits nor to the products they use following screening.

INTERVENTIONS:
Other: Experimental Dentifrice: Stannous Fluoride — Participants will be instructed to dose the toothbrush provided with a strip of dentifrice (a full brush head) on each brushing occasion containing 0.454% w/w Stannous fluoride for 2 minutes twice daily (morning and evening) for 12 weeks.
  Arms: Intervention Group
Device: COREGA Denture Foaming Cleanser — Participant will clean their denture using 2 pumps of the denture cleansing foam and a denture cleaning brush for 90 timed seconds outside of the mouth twice daily (morning and evening) for 12 weeks.
  Arms: Intervention Group
Other: Mouth rinse: Sodium Fluoride — Participants will take 10 ml of the mouth rinse containing 90 ppm sodium fluoride and swished around the mouth for 1 minute twice daily (morning and evening) for 12 weeks.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to investigate the effectiveness of usage of a range of oral products (toothpaste, mouth rinse, denture cleanser) on the oral health of partial denture wearers compared to existing oral hygiene habits.The hypothesis is that there is no treatment difference in the oral health when using the range of products for 12 weeks compared to no intervention.

DETAILED DESCRIPTION:
This study is a single-center, single-blind (to the examiner(s) performing the plaque, gingivitis, denture cleanliness and oral hygiene assessments), randomized, stratified (by denture material type and baseline mean overall modified gingival index [MGI] score), two-treatment, parallel group, 12 week clinical study in generally healthy, adult participants with at least one conventional removable partial denture (RPD) and generalized, mild-moderate, plaque-induced gingivitis (as determined by clinical examiner) and greater than or equal to >=4 natural teeth in each arch that meet all study criteria at both the Screening and Baseline visits (including >= 30 evaluable surfaces for clinical evaluation of gingivitis and plaque). The study will examine the effects of twice daily use of a range of dental/denture products (comprising use of a dentifrice, a mouthrinse and a denture cleanser) compared to no intervention (participants who continue with their existing oral hygiene habits). There will be four visits to the study site: screening, baseline (when participants are randomized), and after 6- and 12 weeks use of the range of dental/denture products.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* A participant with good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant or relevant abnormalities in medical history or upon oral examination, or a condition, that would impact the participant's safety, well being or the outcome of the study, if they were to participate in the study.
* A participant who is a cell phone owner with text messaging capabilities.
* Dental Criteria:

  1. A participant with a minimum of 4 natural teeth in each arch.
  2. A participant with a minimum of 30 scorable surfaces for MGI (Modified Gingival Index), BI (Bleeding Index), OHI (oral hygiene index) and TPI (Turesky Plaque Index). (A scorable surface is defined as a surface that has at least 2/3 of the surface gradable for each clinical index. Third molars, orthodontically banded/bonded, fully crowned or extensively restored or grossly carious teeth are not included in the tooth or scorable surface count. Third molars can be included if, as a result tooth loss, they are functioning as second molars. Tooth surfaces with calculus deposits which, in the opinion of the clinical examiner, would interfere with the assessments of the selected clinical indices are also excluded.)
  3. A participant with a minimum of 2 scorable abutment teeth, defined as teeth proximal to the RPD (removable partial denture) or impinged by an RPD clasp or rest.
  4. A participant with generalized mild-moderate plaque-induced gingivitis present at the screening visit (in the opinion of the clinical examiner from a gross visual examination).
  5. A participant with a mean whole mouth BI >= (greater than or equal to) 0.1 to =< (less than or equal to) 1.3, a mean whole mouth MGI >= 1.75 to =< 2.30 and a mean overall TPI score > (greater than) 1.5 at the Baseline visit.
  6. A participant who habitually wears one conventional removable partial denture constructed of acrylic or cobalt chrome which is acceptable according to the well made and well-fit assessments.

Exclusion Criteria:

* A Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH (GlaxoSmithKline Consumer Healthcare) employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with an acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* A participant who is pregnant (self-reported) or intending to become pregnant over the duration of the study.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who smokes (defined as having smoked or used nicotine products (including ecigarettes, chewing tobacco, gutkha, pan- containing tobacco, nicotine replacement therapies) during the previous 12 months).
* A participant who is unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* A participant with a recent history (within the last year) of alcohol or other substance (e.g. illicit drug) abuse.
* A participant who has previously been enrolled in this study.
* A participant who, in the opinion of the investigator, should not participate in the study.
* Medication Exclusions:

  1. A participant who has taken or is currently taking antibiotics at the Screening visit or in the 14-day period prior to the Baseline visit or requiring antibiotic use prior to dental prophylaxis or other dental procedure.
  2. A participant who is currently taking, on a regular daily basis, an anti-inflammatory, anticoagulant or any other systemic medication (e.g. calcium channel blockers, aspirin therapy, ibuprofen, warfarin) or has a medical condition which, in the opinion of the Investigator, could affect the gingival condition.
  3. A participant who has used an antibacterial mouth rinse (e.g. chlorhexidine, Listerine), dentifrice (e.g. stannous fluoride) or use of any oral care product that, in the opinion of the investigator, could interfere with plaque accumulation or clinical measures within 28 days preceding the baseline visit.
* Oral and Dental Exclusions

  1. A participant with a condition or who is taking medication which, in the opinion of the investigator is causing xerostomia.
  2. A participant who, in the opinion of the investigator, has a periodontal condition that could be adversely affected by lack of immediate periodontal intervention.
  3. A participant who has received treatment for periodontal disease within 12 months of Screening and/or scaling or root surface debridement within 3 months of Screening, which, in the opinion of the Investigator, could compromise study outcomes or the oral health of the participant if they were to participate in the study.
  4. A participant who has numerous restorations in a poor state of repair.
  5. A participant with a severe oral condition (e.g. acute necrotizing ulcerative gingivitis, severe active caries) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they were to participate in the study.
  6. A participant who has had tooth bleaching treatment or a dental prophylaxis within 4 weeks of screening.
  7. A participant who frequently use commercially-available denture cleansers, e.g. denture cleanser tablets, denture cleaning pastes (defined as those participants who use a commercially available cleanser more frequently than once per month).
  8. A participant who currently use denture adhesives (defined as those participants who have used an adhesive in the 28 day period prior to baseline).
  9. A participant who displays evidence of dental fluorosis that might interfere with clinical assessments, as determined by the investigator.
  10. A participant with gingivitis which, in the opinion of the investigator, is not expected to respond to treatment with an over-the-counter dentifrice.
  11. A participant who has an overdenture or orthodontic appliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center in the United Kingdom (UK).
Pre-assignment Details: A total of 61 participants were screened for entry into the study, of whom 58 were enrolled and 49 were randomized to a treatment (24 participants in the intervention group and 25 participants in the non-intervention group) and 48 participants completed the study.
Groups:
- Intervention Group: Participants were instructed to use a dentifrice containing 0.454 percent (%) weight/weight (w/w) stannous fluoride, COREGA denture foaming cleanser and mouth rinse containing 90 parts per million (ppm) sodium fluoride. Participants brushed with a strip of the dentifrice (full brush head) applied to the full length of the toothbrush head for 2 minutes followed by 2 pumps of denture cleanser foam brushed onto removable partial denture (RPD) for 90 seconds and 10 milliliters (ml) of mouth rinse for swished around the mouth for 1 minute. Participants applied all these products topically orally twice daily (morning and evening) for 12 weeks.
- Non-intervention Group: Participants did not receive any products and continued with their existing dental/denture hygiene practices and were instructed not to make changes to either their established habits or to the products they use following screening.
Period: Overall Study
Arm/Group | Intervention Group | Non-intervention Group
Started | 24 | 25
Completed | 23 | 25
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The modified intent to treat (mITT) population was defined as those participants who were randomized, receive at least one dose of study product and had at least one post-baseline efficacy measurement performed.
Groups:
- Intervention Group: Participants were instructed to use a dentifrice containing 0.454% w/w stannous fluoride, COREGA denture foaming cleanser and mouth rinse containing 90 ppm sodium fluoride. Participants brushed with a strip of the dentifrice (full brush head) applied to the full length of the toothbrush head for 2 minutes followed by 2 pumps of denture cleanser foam brushed onto RPD for 90 seconds and 10 ml of mouth rinse for swished around the mouth for 1 minute. Participants applied all these products topically orally twice daily (morning and evening) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Non-intervention Group | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (9.68) | 60.5 (10.30) | 60.4 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 12 | 11 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 2 | 1 | 3
  Asian - Central/South Asian Heritage | 2 | 1 | 3
  Asian - East Asian Heritage | 0 | 1 | 1
  Asian - South East Asian Heritage | 0 | 2 | 2
  White - White/Caucasian/European Heritage | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Bleeding Index (BI) at Week 12
Description: The BI assesses the number of bleeding points elicited on probing as a measure of gingival condition. To perform the assessment, a probe was inserted into the gingival crevice to a depth of approximately 1 millimeter [mm] and then run around the tooth (at approximately 60 degrees to the long axis of the tooth) gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. Three scores were recorded bucally/labially (distal, body, mesial sites) and 3 scores lingually/palatally (distal, body, mesial sites). All scorable teeth in 1 quadrant were probed first (approximately 30 seconds) before recording the number of gingival units which bled. The BI scoring included 3-point scale ranged from 0 to 2, where 0=no bleeding, 1=bleeding within 30 seconds of probing, 2=bleeding immediately on probing. Sites with a score of 1 or 2 were classified as 'bleeding' sites. Higher score indicates worst outcome.
Time Frame: Week 12
Population: mITT Population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Score on a scale | 0.45 (0.036) | 0.76 (0.034)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.40 to -0.20], Standard Error of Mean 0.050

2. Secondary Outcome: Mean Number of Bleeding Sites (NBS) at Week 6 and Week 12
Description: Number of gingival bleeding sites were measured during BI assessment. BI assesses the severity and number of bleeding points elicited on probing as a measure of gingival condition. To perform the assessment, a probe was inserted approximately 1 mm into the gingival sulcus (at approximately 60 degrees) and moved around the tooth, from the distal interproximal area to the mesial interproximal area, gently stretching the gingival epithelium. Sites which showed signs of bleeding immediately on probing or within 30 seconds of probing were classified as a bleeding sites.
Time Frame: Week 6 and Week 12
Population: mITT Population.
Measure: Mean (Standard Error); unit: Number of sites
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Number of sites
  Week 6 | 53.1 (3.40) | 81.7 (3.26)
  Week 12 | 52.9 (3.65) | 80.8 (3.50)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; At Week 6; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -28.6, 95% CI 2-sided [-38.1 to -19.1], Standard Error of Mean 4.73
Statistical Analysis 2: Comparison: Intervention Group vs Non-intervention Group; At Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -27.9, 95% CI 2-sided [-38.2 to -17.7], Standard Error of Mean 5.08

3. Secondary Outcome: Mean Modified Gingival Index (MGI) at Week 6 and Week 12
Description: The MGI focuses on the visual symptoms of gingivitis (redness, texture, edema). The MGI was assessed for the facial and lingual/palatal gingiva of all evaluable teeth, four sites per tooth (facial surface - papilla and margin; lingual/palatal surface - papilla and margin). The MGI scoring included 5-point scale ranged from 0 to 4, where 0=Absence of inflammation, 1=Mild inflammation: slight change in color, little change in texture of any portion of the marginal or papillary gingival unit, 2=Mild inflammation: criteria as (1) but involving the entire marginal or papillary gingival unit, 3=Moderate inflammation: glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit, 4=Severe inflammation: marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Higher score indicates worst outcome.
Time Frame: Week 6 and Week 12
Population: mITT Population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Score on a scale
  Week 6 | 1.52 (0.044) | 1.92 (0.043)
  Week 12 | 1.50 (0.039) | 1.86 (0.038)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; At Week 6; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.52 to -0.27], Standard Error of Mean 0.062
Statistical Analysis 2: Comparison: Intervention Group vs Non-intervention Group; At Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.47 to -0.25], Standard Error of Mean 0.054

4. Secondary Outcome: Mean Overall Turesky Plaque Index (TPI) at Week 6 and Week 12
Description: Supra-gingival plaque was assessed on the facial and lingual/palatal surfaces of all scorable teeth, six sites per tooth using TPI which indicated plaque accumulation in the gingival area of the tooth. Each tooth surface was divided into 3 areas; three scores were recorded facially (mesiofacial, facial, distofacial) and three scores lingually (mesiolin-gual, lingual and distolingual) generating a total of six scores per tooth. The plaque was disclosed and scored on a 6-point scale ranged from 0 to 5 where: 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin, 3=Band of plaque wider than 1 mm but covering less than (<) 1/3 of the tooth surface, 4=Plaque covering greater than or equal to (>=) 1/3 but < 2/3 of the tooth surface, 5=Plaque covering >= 2/3 of the tooth surface. Higher score indicates worst outcome.
Time Frame: Week 6 and Week 12
Population: mITT Population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Score on a scale
  Week 6 | 2.12 (0.102) | 2.97 (0.098)
  Week 12 | 2.07 (0.100) | 3.02 (0.096)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; At Week 6; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.14 to -0.56], Standard Error of Mean 0.142
Statistical Analysis 2: Comparison: Intervention Group vs Non-intervention Group; At Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.23 to -0.67], Standard Error of Mean 0.139

5. Secondary Outcome: Mean Interproximal TPI at Week 6 and Week 12
Description: Supra-gingival plaque was assessed on the facial and lingual/palatal surfaces of all scorable teeth, six sites per tooth using TPI which indicated plaque accumulation in the gingival area of the tooth. Each tooth surface was divided into 3 areas; three scores were recorded facially (mesiofacial, facial, distofacial) and three scores lingually (mesiolin-gual, lingual and distolingual) generating a total of six scores per tooth. The plaque was disclosed and scored on a 6-point scale ranging from 0 to 5, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin, 3=Band of plaque wider than 1 mm but covering < 1/3 of the tooth surface, 4=Plaque covering >= 1/3 but < 2/3 of the tooth surface, 5=Plaque covering >= 2/3 of the tooth surface. Higher score indicates worst outcome.
Time Frame: Week 6 and Week 12
Population: mITT Population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Score on a scale
  Week 6 | 2.31 (0.108) | 3.22 (0.104)
  Week 12 | 2.24 (0.111) | 3.29 (0.106)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; At Week 6; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.22 to -0.61], Standard Error of Mean 0.151
Statistical Analysis 2: Comparison: Intervention Group vs Non-intervention Group; At Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.36 to -0.74], Standard Error of Mean 0.154

6. Secondary Outcome: Mean BI at Week 6
Description: The BI assesses the number of bleeding points elicited on probing as a measure of gingival condition. To perform the assessment, a probe was inserted into the gingival crevice to a depth of approximately 1 mm and then run around the tooth (at approximately 60 degrees to the long axis of the tooth) gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. Three scores were recorded bucally/labially (distal, body, mesial sites) and 3 scores lingually/palatally (distal, body, mesial sites). All scorable teeth in 1 quadrant were probed first (approximately 30 seconds) before recording the number of gingival units which bled. The BI scoring included 3-point scale ranged from 0 to 2, where 0=no bleeding, 1=bleeding within 30 seconds of probing, 2=bleeding immediately on probing. Sites with a score of 1 or 2 were classified as 'bleeding' sites. Higher score indicates worst outcome.
Time Frame: Week 6
Population: mITT Population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Score on a scale | 0.45 (0.033) | 0.76 (0.031)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.41 to -0.23], Standard Error of Mean 0.045

7. Secondary Outcome: Mean Partial Denture Cleanliness Index (PDCI) at Week 6 and 12
Description: The cleanliness of the partial denture was evaluated based on the modification of the Clinical Categorization of Denture Cleanliness Index. A suitable dental probe was used to gently scrape the surfaces of the RPD and the PDCI was scored. All surfaces of the RPD were assessed and the highest score applicable was recorded. PDCI scoring system included 5-point scale ranged from 0 to 4, where 0=No visible plaque; no matter adherent to the dental probe on light scraping, 1=No visible plaque; matter adherent to the dental probe on light scraping, 2=Deposits of plaque just visible on careful examination without need to confirm by scraping, 3=Deposits of plaque clearly visible, 4=Gross plaque deposits ("velvet appearance"). Higher score indicates worst outcome.
Time Frame: Week 6 and Week 12
Population: mITT Population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Score on a scale
  Week 6 | 1.2 (0.12) | 1.7 (0.12)
  Week 12 | 1.1 (0.11) | 1.9 (0.10)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; At Week 6; Test type: Superiority; p = 0.0039, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.9 to -0.2], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Intervention Group vs Non-intervention Group; At Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.1 to -0.5], Standard Error of Mean 0.15

8. Secondary Outcome: Mean Calculus Index (CI) at Week 6 and Week 12
Description: The extent of calculus on each tooth surface (buccal and lingual) was determined by visual examination. Only definite deposits of hard calculus were recorded. The CI was assessed on the facial and lingual surfaces of each scorable tooth. The CI for each participant was calculated as the mean score of all tooth surfaces (facial/lingual). CI scoring included 4-point scale ranged from 0 to 3 where: 0=No calculus present, 1=Supragingival calculus covering not greater than (>) 1/3 of exposed tooth surface, 2=Supragingival calculus covering > 1/3 but not > 2/3 of exposed tooth surface or presence of individual flecks of Subgingival calculus around cervical portion of tooth or both, 3= supragingival calculus covering > 2/3 of exposed tooth surface or a continuous band of Subgingival calculus around cervical portion of tooth or both. Higher score indicates worst outcome.
Time Frame: Week 6 and Week 12
Population: mITT Population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Score on a scale
  Week 6 | 0.08 (0.036) | 0.19 (0.034)
  Week 12 | 0.10 (0.024) | 0.18 (0.023)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; At Week 6; Test type: Superiority; p = 0.0367, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.21 to -0.01], Standard Error of Mean 0.050
Statistical Analysis 2: Comparison: Intervention Group vs Non-intervention Group; At Week 12; Test type: Superiority; p = 0.0725, Van-Elteren test; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.14 to -0.01], Standard Error of Mean 0.033

9. Secondary Outcome: Mean Oral Debris Index (ODI) at Week 6 and Week 12
Description: The extent of oral debris (defined as soft foreign matter on the surface of teeth) on each tooth surface was determined by running the side of a number 5 explorer (Shephard's crook) probe along the buccal, labial and lingual surfaces and noting the occlusal or incisal extent of the debris as it was removed from the tooth surface. The ODI was assessed on the facial and lingual surfaces of each scorable tooth. The ODI for each participant was calculated as the mean score of all tooth surfaces (facial/lingual).ODI scoring system included 4-point scale ranged from 0 to 3 where: 0=No debris or stain present, 1=Soft debris covering not > 1/3 of the tooth surface the presence of extrinsic stains without other debris regardless of surface area covered, 2= Soft debris covering more than one third, but not more than two thirds, of the exposed tooth surface, 3=Soft debris covering more than two thirds of the exposed tooth surface. Higher score indicates worst outcome.
Time Frame: Week 6 and Week 12
Population: mITT Population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Score on a scale
  Week 6 | 0.22 (0.054) | 0.50 (0.052)
  Week 12 | 0.20 (0.052) | 0.46 (0.050)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; At Week 6; Test type: Superiority; p = 0.0006, ANCOVA; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.43 to -0.13], Standard Error of Mean 0.075
Statistical Analysis 2: Comparison: Intervention Group vs Non-intervention Group; At Week 12; Test type: Superiority; p = 0.0009, ANCOVA; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.41 to -0.11], Standard Error of Mean 0.073

10. Secondary Outcome: Mean Oral Hygiene Index (OHI) at Week 6 and Week 12
Description: OHI was calculated as sum score of mean CI and mean ODI. CI scoring:0=no calculus present,1=supragingival calculus covering not >1/3 of exposed tooth surface,2=supragingival calculus covering >1/3 but not >2/3 of exposed tooth surface/presence of individual flecks of subgingival calculus around cervical portion of tooth/both,3=supragingival calculus covering >2/3 of exposed tooth surface/continuous band of subgingival calculus around cervical portion of tooth/both. ODI scoring:0=no debris/stain present,1= supragingival calculus covering not >1/3 of exposed tooth surface,2=supragingival calculus covering>1/3 but not >2/3 of exposed tooth surface/presence of individual flecks of subgingival calculus around cervical portion of tooth/both,3=supragingival calculus covering >2/3 of exposed tooth surface/continuous band of subgingival calculus around cervical portion of tooth/ both. Thus, total OHI score range was 0 to 6. Higher score indicates worst outcome.
Time Frame: Week 6 and Week 12
Population: mITT Population.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 23 | 25
Score on a scale
  Week 6 | 0.30 (0.085) | 0.69 (0.081)
  Week 12 | 0.30 (0.065) | 0.64 (0.062)
Statistical Analysis 1: Comparison: Intervention Group vs Non-intervention Group; At Week 6; Test type: Superiority; p = 0.0020, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.62 to -0.15], Standard Error of Mean 0.117
Statistical Analysis 2: Comparison: Intervention Group vs Non-intervention Group; At Week 12; Test type: Superiority; p = 0.0005, ANCOVA; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.52 to -0.16], Standard Error of Mean 0.090

ADVERSE EVENTS:
Time Frame: All adverse events (AEs), and therefore all serious AEs (SAEs) were collected immediately after a participant consent to participate in the study until 5 days following last administration of the study product (or last procedure) (Up to Week12).
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study product including any washout or lead-in product (or medical device). A SAE is a particular category of an adverse event where the adverse outcome is serious.
Arm/Group | Intervention Group | Non-intervention Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 3/24 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=24) | Non-intervention Group (N=25)
COVID-19 (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Burn oral cavity (Injury, poisoning and procedural complications) | 1 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT04290624/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT04290624/SAP_001.pdf